CLINICAL TRIAL: NCT07307469
Title: Compassionate Administration of ZVS101e Injection for Extended Treatment
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chigenovo Co., Ltd (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZYA-2025-004
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Patients With Bietti Crystalline Corneoretinal Dystrophy (Carrying Biallelic CYP4V2 Mutations)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Safety evaluation (Experimental): Adverse events that occurred during the study period
  Interventions: Drug: ZVS101e

INTERVENTIONS:
Drug: ZVS101e — ZVS101e is a recombinant adeno-associated virus serotype 8 (rAAV8) vector expressing human CYP4V2 protein

SUMMARY:
To provide treatment options for the control group of subjects who completed the 52-week follow-up of the Phase III clinical trial (Protocol number: ZYA-2024-001) of ZVS101e in subjects with crystalline retinal degeneration (BCD).

DETAILED DESCRIPTION:
The trial period lasts for a total of 8 weeks, including a 4-week screening period, a administration period, and visits on the 1st day, 7th day, and 4th week after administration. The patients were followed up at the research center on the 1st day, 7th day and 4th week after administration to evaluate the safety.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who were randomly assigned as the control group in a multicenter, randomized controlled, Phase III clinical trial (Protocol number: ZYA-2024-001) on the efficacy and safety of a single subretinal injection of ZVS101e in subjects with crystalline retinal degeneration (BCD) and completed a 52-week safety follow-up were included.
2. Voluntarily participate in clinical trials and sign informed consent forms, and be willing to complete all trial procedures as required by the protocol.
3. Study the BCVA of the eye ≤60 ETDRS letters.

Exclusion Criteria:

1. The study eye currently has or has had macular degeneration such as macular holes or neovascularization in the macular area; Other ocular diseases such as glaucoma and diabetic retinopathy that may hinder surgery or interfere with the interpretation of the study endpoint.
2. The study eye had undergone retinal repositioning surgery, vitrectomy, or had undergone any intraocular surgery within 3 months prior to enrollment, such as phacoemulsification for cataract.
3. Within one month prior to enrollment, the patient had a viral infectious disease that may affect the efficacy and safety evaluation of the investigational drug or had received an antiviral vaccine.
4. Any eye has previously received gene therapy or stem cell therapy for BCD and other ocular diseases, including but not limited to other viral vector gene therapies, mRNA therapies, etc.
5. Known to be allergic to the drugs planned to be used in the study.
6. The following laboratory test abnormalities have clinical significance:

   Liver function: ALT or AST>2 times the upper limit of the normal value; Abnormal coagulation function (prothrombin time ≥ the upper limit of normal value by 3 seconds, activated partial thromboplastin time ≥ the upper limit of normal value by 10 seconds).
7. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation | 4 weeks
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No